CLINICAL TRIAL: NCT04127435
Title: Clinical Study on Pelvic Recurrence of Gynecologic Tumors After External Irradiation by Three Dimensional Printing Personalized Template Assisted With 192Ir High Dose Rate Interstitial Brachytherapy
Brief Title: High Dose Rate Interstitial Brachytherapy With Three Dimensional Printing Template for Recurrent Gynecologic Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019338-1
Record Dates: First submitted 2019-09-01; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-Dose-Rate 192Ir Brachytherapy: 1. All patients underwent computed tomography (CT) 3-5 days before surgery. The collimation is 2.5 mm and CT Planning System.
  2. Delineation of the gross tumor volume (GTV) and adjacent organs at risk (OARs);
  3. Determination of the needle tract of the implanted insertion direction, distribution, and depth. Then calculation of the dose distribution of the target volume and OARs.
  4. Depending on B-TPS data, we establish a digital model for the individual template.
  5. Local anesthesia or intraspinal anesthesia was induced in all patients. The three-dimensional printing noncoplanar templates (3D-PNCT) was placed on the surface of the treatment area of the patient. The 3D-PNCT was aligned accurately with the outer-contour features. Through the guide hole of the 3D-PNCT, we inserted to pre-planned depths.
  6. Delineation of the GTV and design planning .
  7. Connect the source tube and 192Ir high dose rate interorganizational brinotherapy
  8. At the end pressed to stop bleeding.

SUMMARY:
This is a single-center study.Eligible patients will have histologically proven pelvic recurrence of cervical cancer after radiotherapy .

DETAILED DESCRIPTION:
The results of treatment, examination and follow-up of patients with recurrent cervical cancer after radiotherapy who recieved imaging guided three dimensional printing personalized template assisted with 192Ir high dose rate interorganizational braided therapy were statistically analyzed .

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed pelvic recurrence of cervical cancer.
* Age ≥ 18 years and ≤ 75 years.
* Previous accept pelvic radiotherapy;
* Karnofsky ≥60；
* Patients reject or cannot tolerate surgery;
* Received 192Ir high dose rate intertissue salvage therapy;
* Ultrasound guidance or computed tomography guidance;
* Regular review and follow-up.

Exclusion Criteria:

* Patients participated in clinical trials of other drugs within four weeks;
* The patient had a previous history of bleeding, and any bleeding event with severity rating of CTCAE5.0 or above occurred within 4 weeks prior to screening;
* There are any puncture taboos.
* Patients with severe cardiovascular and cerebrovascular diseases.
* Unable to treat as planned.
* Patients lack major indicators and cannot participate in post-treatment review and follow-up.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed pelvic recurrence of cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Progression Free Survival | 2 years
  Local progression free survival was defined as the time from the implantation of the treatment to the treatment of local tumor progression.
Tumor Response Rate | three months
  Tumor size changes were monitored using CT. According to the solid tumor treatment efficacy evaluation standard RECIST, evaluation results including complete response, partial response, stable disease, and progression disease.Tumor response rate was complete response rate plus partial response rate.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival was defined as the time from the implantation of the treatment to the death of any cause.
Safety and Tolerability | 2 years
  Number of participants with treatment-related acute adverse events were evaluated according to RTOG acute radiation injury grading standards; Number of participants with treatment-related late adverse events were evaluated according to RTOG/ EORTC advanced radiation injury grading schemes.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jiang, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Peking University Third Hospital, Beijing, China